CLINICAL TRIAL: NCT05570929
Title: Observation of Alterations in Kidney Function, Immune System and Gut Mircobiota After Living Donor Kidney Transplantation
Brief Title: LONGitudinal Multi-omics Phenotyping of KIDney Function Alteration
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Till Schütte, Principle Investigator, Charite University, Berlin, Germany
Other Study IDs: LONGKID
Record Dates: First submitted 2022-09-28; First posted 2022-10-07 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Chronic Kidney Diseases
Keywords: Short chain fatty acids; Shannon-Index; Microbial diversity; Home sampling; Kidney transplant
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, urine, stool, and peripheral blood mononuclear cells will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kidney Donor: Defined as a human individual donating a kidney
- Kidney Recipient: Defined as a patient suffering from chronic kidney disease being the recipient of a kidney transplant

SUMMARY:
This is a longitudinal observation of kidney function, immune system and gut microbiota before and 24 weeks after a live kidney transplantation conducted in donor and recipient pairs living in the same household. Outcome measures include kidney function, body composition, blood pressure, gut microbiome composition, metabolomics and immune cell states.

ELIGIBILITY:
Inclusion Criteria:

* Body-Mass-Index 18,5 - 34,9 kg/m2
* Planned living kidney donation / transplantation

Exclusion Criteria:

* Clinically relevant heart, lung, liver, and kidney diseases
* Postoperative phase
* Acute infections
* Vegan diet
* Change of body weight of more than 10% in the month prior to study entry
* Known drug or alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Fecal microbiome taxonomy (Shannon-Index) | Change from Baseline at 24 weeks
  Measured by 16S amplicon sequencing

SECONDARY OUTCOMES:
Functional capacity of gut microbiota | Change from Baseline at 24 weeks
  Measured by metagenome sequencing
Frequency of circulating T-cell subtypes | Change from Baseline at 24 weeks
  Measured by flow cytometry (%)
Serum tryptophan metabolites concentration | Change from Baseline at 24 weeks
  Measured by mass spectrometry
Serum short-chain fatty acid concentration | Change from Baseline at 24 weeks
  Measured by mass spectrometry
Fecal tryptophan metabolites concentration | Change from Baseline at 24 weeks
  Measured by mass spectrometry
Fecal short-chain fatty acid concentration | Change from Baseline at 24 weeks
  Measured by mass spectrometry
Office systolic blood pressure | Change from Baseline at 24 weeks
  Mean of five consecutive blood pressure measurements (mmHg)
Office diastolic blood pressure | Change from Baseline at 24 weeks
  Mean of five consecutive blood pressure measurements (mmHg)
Body fat content | Change from Baseline at 24 weeks
  Measured by bioelectrical impedance analysis (%)
Fat free mass | Change from Baseline at 24 weeks
  Measured by bioelectrical impedance analysis (%)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Wilck, MD, Principal Investigator — Charite University, Berlin, Germany; Hendrik Bartolomaeus, MD, Principal Investigator — Charite University, Berlin, Germany; Anja Mähler, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Experimental and Clinical Research Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of reported articles (text, tables, figures, supplemental data) will be shared after deidentification.
Time Frame: Beginning in 2 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.